CLINICAL TRIAL: NCT01107080
Title: Fast Spectral Imaging Device for Tumor Margin Mapping
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00017428; 2R42CA128160-02 (NIH)
Record Dates: First submitted 2010-04-18; First posted 2010-04-20 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast carcinoma in situ; ductal breast carcinoma in situ; invasive carcinoma; invasive ductal carcinoma; invasive lobular carcinoma
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Lobular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Degradation: 30 mastectomy, partial mastectomy, and mammoplasty samples will be analyzed to define the effective post-excision time window in which the device must be used before the results can no longer be evaluated. The mammoplasty specimens are necessary to assess normal tissue outcomes.
- Reproducibility: 25 Partial Mastectomy cases will be analyzed to distinguish between different implementation methods of the technology.

SUMMARY:
The objective of the proposed research is to develop a clinical-trial-ready device and to evaluate its practical utility as a routinely used intra-operative tool. Our multidisciplinary group has previously shown that optical techniques can effectively discriminate between malignant and non-malignant breast tissues. The proposed technology will be a multi-channel optical assay device for intra-operative imaging of margins in specimens excised from patients undergoing breast conserving surgery (partial mastectomy) or mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a partial mastectomy or mastectomy for the treatment of an invasive or non-invasive breast malignancy
* Age > 18
* Clinically detectable disease either by physical examination or radiographic studies
* Patients of all ethnic and gender groups will be included. Protocol accrual will be reviewed annually to include a determination of minority and gender representation. If accrual demonstrates under representation of any group with comparison to disease incidence in that group, appropriate measures will be undertaken to increase participation of patients of that minority or gender group.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients considered in "vulnerable" populations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 2 groups of patients and each group contains 20 participants.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To perform a critical evaluation of the device in a practical clinical setting | 2 years
  (1) In order to define the effective post-excision time window in which the device must be used, which ultimately has bearings on the final product indications for use. (2)To analyze the different methods of implementation of the technology.

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi Ramanujam, PhD, Study Chair — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States